CLINICAL TRIAL: NCT03581240
Title: An Intermediate Expanded Use Trial of DFMO
Status: Available | Type: Expanded Access
Sponsor: Giselle Sholler (Other)
Collaborators: K C Pharmaceuticals Inc. (Industry); USWM, LLC (Unknown)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Study Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Other Study IDs: NMTRC006
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Neuroblastoma; Medulloblastoma; Typical Teratoid Rhabdoid Tumor; Embryonal Tumor With Abundant Neuropil and True Rosettes; Ependymoblastoma; Medulloepithelioma
MeSH Terms: conditions — Neuroblastoma; Medulloblastoma; Typical Teratoid Rhabdoid Tumor; Neuroectodermal Tumors, Primitive | interventions — Eflornithine

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: eflornithine HCl — In this study subjects without CNS disease will receive oral difluoromethylornithine (DFMO) at a dose of 500 to 1000 mg/m2 BID
  Subjects with CNS disease will receive a dose of 2500 mg/m2/dose BID in order to facilitate crossing into the CNS.
  Other Names: DFMO

SUMMARY:
To provide DFMO in an expanded use setting to subjects with relapsed rare tumors with increased LIN28 expression or MYCN amplification or up regulation of ornithine decarboxylase.

ELIGIBILITY:
Inclusion Criteria:

* Age: 0-30 years at the time of initial diagnosis.
* Diagnosis: Histologic verification at either the time of original diagnosis or a previous relapse of High Risk neuroblastoma, medulloblastoma, atypical teratoid rhabdoid tumor, embryonal tumor with abundant neuropil and true rosettes, ependymoblastoma, medulloepithelioma and other rare pediatric MYC, ODC or LIN28/Let7 driven tumors (each type will form a new subset).
* Disease Status: Subjects must be in one of the following disease categories:

  1. High risk neuroblastoma patients that have completed standard of care upfront therapy and are not eligible for NMTRC014.
  2. Medulloblastoma patients who have completed standard of care therapies.
  3. Relapsed/refractory neuroblastoma patients who have completed standard of care therapies.
  4. Rare tumors with increased LIN28 expression or MYCN amplification or up regulation of ornithine decarboxylase who have completed standard of care therapies.
* Subjects are not eligible to enroll on DFMO studies NMTRC002, NMTRC003, NMTRC010, or NMTRC014.
* A negative serum or urine pregnancy test is required for female subjects of child bearing potential (onset of menses or ≥13 years of age).
* Both male and female post-pubertal study subjects need to agree to use one of the more effective birth control methods during treatment and for six months after treatment is stopped. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonorgestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended.
* Informed Consent: All subjects and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* BSA (m2) of <0.25
* Investigational Drugs: Subjects who are currently receiving another investigational drug are excluded from participation.

Ages: 0 Years to 30 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — Beat Childhood Cancer
Locations (1):
- Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania, United States

REFERENCES:
- See also: Beat Childhood Cancer website — http://beatcc.org